CLINICAL TRIAL: NCT03895489
Title: Comparative Effectiveness of the Journey Total Knee Arthroplasty Relative to Two Standard of Care Total Knee Arthroplasty Prostheses: A Randomized Controlled Trial
Brief Title: Effectiveness of the Journey Total Knee Arthroplasty Versus Two Standard of Care Total Knee Arthroplasty Prostheses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00087023
Record Dates: First submitted 2019-01-29; First posted 2019-03-29 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Journey II (Experimental): Smith and Nephew Richards (SNR) Journey II Knee prosthesis
  Interventions: Device: Journey II
- Stryker (Active Comparator): Stryker Triathlon Total Knee prosthesis
  Interventions: Device: Stryker
- Zimmer (Active Comparator): Zimmer Persona® The Personalized Knee prosthesis
  Interventions: Device: Zimmer

INTERVENTIONS:
Device: Journey II — Smith and Nephew Richards (SNR) Journey II Knee prosthesis
  Arms: Journey II
Device: Stryker — Stryker Triathlon Total Knee prosthesis
  Arms: Stryker
Device: Zimmer — Zimmer Persona® The Personalized Knee prosthesis
  Arms: Zimmer

SUMMARY:
The purpose of the study is to determine if knee replacement performed using Journey II implant is different from two other standard-of-care knee replacements using Stryker and Zimmer in terms of knee movements and forces, walking patterns, pain, and function after surgery.

DETAILED DESCRIPTION:
Background

Osteoarthritis is the most prevalent form of arthritis, with weight-bearing joints, particularly the knee commonly affected. Osteoarthritis is a leading cause of mobility disability and is associated with functional loss in adults. Total knee arthroplasty (TKA) is cost-effective and successful for those with end-stage knee osteoarthritis. In 2016/17, about 67,169 TKAs were performed in Canada, an increase of 16% since 2012/13.

Justification

TKA aims to improve joint mechanics as well as knee pain and function. Patients indicate that their primary expectations following TKA are improved pain and walking ability. Most TKA implants are fixed bearing (such as Stryker and Zimmer) with no movement of the implant with knee motion. The Journey II TKA has a medial pivot function that may improve patient outcomes further, by replicating meniscal function. However, this has not yet been proven as it would require more specific measurement of knee kinetics and kinematics such as we propose here.

The outcome of this study will provide information about knee pain, movements (kinematics) and forces (kinetics) and walking patterns after TKA using different implants. Through this study, we should be able to inform future research on rehabilitation protocols to alter knee movements after TKA, while enhancing patients' function and quality of life.

Hypotheses

Primary Hypothesis: We hypothesize that TKA performed using the Smith and Nephew Richards (SNR) Journey II TKA system will be superior to standard TKA prostheses (Stryker Triathlon Total Knee System and Zimmer Persona® The Personalized Knee) in terms of knee biomechanics (knee kinematics and kinetics) and spatio-temporal gait parameters at 1-year post-TKA using the Computer-Assisted Rehabilitation ENvironment (CAREN).

Secondary Hypothesis: We hypothesize that the Smith and Nephew Richards (SNR) Journey II TKA will provide increased improvement from preoperative levels in pain and function in comparison to standard TKA prostheses.

Objectives

Primary Objective: The primary objective of this randomized, comparative trial is to demonstrate that TKA performed using the Smith and Nephew Richards (SNR) Journey II TKA system is superior to standard TKA prostheses (Stryker Triathlon Total Knee System and Zimmer Persona® The Personalized Knee) in terms of knee biomechanics (knee kinematics and kinetics) and spatio-temporal gait parameters at 1-year post-TKA using the Computer-Assisted Rehabilitation ENvironment (CAREN). We will evaluate these parameters for level treadmill walking.

Secondary Objective: The secondary objective of this study will be to demonstrate that the Smith and Nephew Richards (SNR) Journey II TKA provides increased improvement from preoperative levels in pain and function in comparison to standard TKA prostheses. The new Knee Society Clinical Rating Scores (KSCRS) will be calculated preoperatively and at 1 year and 2 years postoperatively with the potential for longer-term follow-up. Patient questionnaires will be assessed preoperatively and at each postoperative interval.

Study Design: A prospective, randomized, post-market, comparative design will be employed.

Participants: A total of 75 participants will be enrolled in this study. Twenty-five (25) participants will receive the Journey II TKA System. Fifty (50) participants will receive standard TKA: 25 will receive the Stryker Triathlon Total Knee System and 25 will receive Zimmer Persona® The Personalized Knee, which are commonly used in this zone.

Randomization: This study will utilize a computer-generated 1:1 randomization scheme. The randomization schedule will be maintained and controlled by Collaborative Orthopaedic REsearch (CORe) at the University of Alberta. The investigators and research associates will not have access to this schedule. When an eligible patient meets the criteria for inclusion in the study and signs the informed consent form, the research associate will open a sequentially-numbered envelope that contains the group allocation. Baseline gait evaluation will be completed for randomized patients. Any deviation from the assigned treatment group will be reported as a deviation from the protocol. Participants deviating from the randomization assignment will continue to be followed, and data collected will be reported as per intention to treat principles.

Estimated Study Duration: The enrollment period is estimated to last a maximum of 18 to 24 months. Participants will be evaluated per the evaluation schedule until the 2 year follow-up time point (secondary objective). It is possible that the study will be extended to longer-term follow-up to evaluate long-term performance.

Pre-operative visit

During the preoperative visit, patients who are possible candidates for this study will be screened to determine if they meet the inclusion/exclusion criteria. If the patient is a candidate, the investigator will propose participation in the study to the patient, and the patient will be given a consent-to-contact form by the investigator. If the patient consents to be contacted, the research associate would contact the patient to provide more details about the study. If the patient is willing to proceed with the study, an approved informed consent form must be signed by the patient prior to participating in any study related activities.

Once the patient has consented to participate in the study, preoperative data will be collected including: demographics, medical history, preoperative gait analysis and functional evaluation (KSCRS), EQ-5D - a standardized instrument that measures health-related quality of life, UCLA activity-level rating (UCLA), knee injury and osteoarthritis outcome score (KOOS), and the Forgotten Joint Score.

Follow-up visits

Gait analysis and patient-reported outcomes (PRO) data will be collected at the following postoperative intervals: 1-year (gait and PRO), 2 years (PRO) and potentially during longer-term follow-up (PRO).

ELIGIBILITY:
Inclusion Criteria:

1. Participant has signed an approved informed consent form.
2. Participant is a male or non-pregnant female and aged 50 to 75 years at the time of study device implantation.
3. Participant has a diagnosis of Non-Inflammatory Degenerative Joint Disease (NIDJD).
4. Participant is a candidate for a primary posterior-stabilized total knee replacement.
5. Participant is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

1. Participant has a Body Mass Index (BMI) ≥ 40 kg/m2.
2. Participant has a varus or valgus deformity greater than 15º or flexion contracture greater than 20º or knee flexion range of motion < 90º in either lower extremity.
3. Participant has an active or suspected latent infection in or about the affected knee joint at time of study device implantation.
4. Participant has received any orthopaedic surgical intervention to the lower extremities within the past 6 months or is expected to require any orthopaedic surgical intervention to the lower extremities, other than the TKA, within the next year.
5. Participant requires bilateral total knee replacements, or has a history of contralateral partial or total knee replacement within the past 6 months.
6. Participant has other medical conditions which limit the ability to evaluate the safety and efficacy of the device.
7. Participant requires revision surgery of a previously implanted total knee replacement or knee fusion to the affected joint.
8. Participant has a known sensitivity to device materials.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-09-09 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
knee flexion-extension range of motion (ROM) during level treadmill walking | 1 month preoperative
  Angle of knee measured using the Computer-Assisted Rehabilitation Environment (CAREN).
  Unit: Degree
knee flexion-extension range of motion (ROM) during level treadmill walking | 1 year post-operative
  Angle of knee measured using the Computer-Assisted Rehabilitation Environment (CAREN).
  Unit: Degree
knee abduction-adduction range of motion (ROM) during level treadmill walking | 1 month preoperative
  Angle of knee measured using the Computer-Assisted Rehabilitation Environment (CAREN).
  Unit: Degree
knee abduction-adduction range of motion (ROM) during level treadmill walking | 1 year post-operative
  Angle of knee measured using the Computer-Assisted Rehabilitation Environment (CAREN).
  Unit: Degree
Max velocity of knee flexion-extension during level treadmill walking | 1 month preoperative
  Knee velocity measured using the Computer-Assisted Rehabilitation Environment (CAREN). Unit: degree/s
Max velocity of knee flexion-extension during level treadmill walking | 1 year post-operative
  Knee velocity measured using the Computer-Assisted Rehabilitation Environment (CAREN). Unit: degree/s
Max velocity of knee abduction-adduction during level treadmill walking | 1 month preoperative
  Knee velocity measured using the Computer-Assisted Rehabilitation Environment (CAREN).
  Unit: degree/s
Max velocity of knee abduction-adduction during level treadmill walking | 1 year post-operative
  Knee velocity measured using the Computer-Assisted Rehabilitation Environment (CAREN).
  Unit: degree/s
Max moment of knee flexion-extension during level treadmill walking | 1 month preoperative
  Knee moment measured using the Computer-Assisted Rehabilitation Environment (CAREN).
  Unit: Newton meter
Max moment of knee flexion-extension during level treadmill walking | 1 year post-operative
  Knee moment measured using the Computer-Assisted Rehabilitation Environment (CAREN).
  Unit: Newton meter
Max moment of knee abduction-adduction during level treadmill walking | 1 month preoperative
  Knee moment measured using the Computer-Assisted Rehabilitation Environment (CAREN).
  Unit: Newton meter
Max moment of knee abduction-adduction during level treadmill walking | 1 year post-operative
  Knee moment measured using the Computer-Assisted Rehabilitation Environment (CAREN).
  Unit: Newton meter

SECONDARY OUTCOMES:
Walking velocity during level treadmill walking | 1 month preoperative
  Walking velocity (the quotient of the distance traveled by the time) measured using the Computer-Assisted Rehabilitation Environment (CAREN).
  Unit: m/s
Walking velocity during level treadmill walking | 1 year post-operative
  Walking velocity (the quotient of the distance traveled by the time) measured using the Computer-Assisted Rehabilitation Environment (CAREN).
  Unit: m/s
Cadence during level treadmill walking | 1 month preoperative
  Cadence (the quotient of the number of steps taken per minute) measured using the Computer-Assisted Rehabilitation Environment (CAREN).
  Unit: Steps/min
Cadence during level treadmill walking | 1 year post-operative
  Cadence (the quotient of the number of steps taken per minute) measured using the Computer-Assisted Rehabilitation Environment (CAREN).
  Unit: Steps/min
Stride length during level treadmill walking | 1 month preoperative
  Stride length (the distance between the position (e.g., heel strike) of one foot to the next similar position in the same foot (e.g. next heel strike)) measured using the Computer-Assisted Rehabilitation Environment (CAREN).
  Unit: meter
Stride length during level treadmill walking | 1 year post-operative
  Stride length (the distance between the position (e.g., heel strike) of one foot to the next similar position in the same foot (e.g. next heel strike)) measured using the Computer-Assisted Rehabilitation Environment (CAREN).
  Unit: meter
The new Knee Society Clinical Rating Scores (KSCRS) | 1 month preoperative
  The function subscale of this scorning system (KSCRS) quantifies the function of the knee.
  Score: 100
The new Knee Society Clinical Rating Scores (KSCRS) | 1 year post-operative
  The function subscale of this scorning system (KSCRS) quantifies the function of the knee.
  Score: 100
The new Knee Society Clinical Rating Scores (KSCRS) | 2 years post-operative
  The function subscale of this scorning system (KSCRS) quantifies the function of the knee.
  Score: 100
Euro-Quality of Life five dimensions questionnaire (EQ-5D) | 1 month preoperative
  Standardized instrument that measures health-related quality of life. consists of 2 parts:
  1. EQ-5D-5L: self-report, generic health utility instrument with 5 domains (mobility, self-care, pain/discomfort, depression/anxiety, and usual activities) and 5 levels in each domain (no problems, slight problems, moderate problems, severe problems, and extreme problems).
  2. EQ Visual Analogue scale (EQ VAS): Scores: 100 = the best health you can imagine and 0 = the worst health you can imagine.
Euro-Quality of Life five dimensions questionnaire (EQ-5D) | 1 year post-operative
  Standardized instrument that measures health-related quality of life. consists of 2 parts:
  1. EQ-5D-5L: self-report, generic health utility instrument with 5 domains (mobility, self-care, pain/discomfort, depression/anxiety, and usual activities) and 5 levels in each domain (no problems, slight problems, moderate problems, severe problems, and extreme problems).
  2. EQ Visual Analogue scale (EQ VAS): Scores: 100 = the best health you can imagine and 0 = the worst health you can imagine.
Euro-Quality of Life five dimensions questionnaire (EQ-5D) | 2 years post-operative
  Standardized instrument that measures health-related quality of life. consists of 2 parts:
  1. EQ-5D-5L: self-report, generic health utility instrument with 5 domains (mobility, self-care, pain/discomfort, depression/anxiety, and usual activities) and 5 levels in each domain (no problems, slight problems, moderate problems, severe problems, and extreme problems).
  2. EQ Visual Analogue scale (EQ VAS): Scores: 100 = the best health you can imagine and 0 = the worst health you can imagine.
UCLA activity-level rating (UCLA) | 1 month preoperative
  Scale to assess activity ranging from 1 to 10. The patient indicates her or his most appropriate activity level, with 1 defined as ''wholly inactive and dependent on others'' and 10 defined as ''regular participation in impact sports.''
UCLA activity-level rating (UCLA) | 1 year post-operative
  Scale to assess activity ranging from 1 to 10. The patient indicates her or his most appropriate activity level, with 1 defined as ''wholly inactive and dependent on others'' and 10 defined as ''regular participation in impact sports.''
UCLA activity-level rating (UCLA) | 2 years post-operative
  Scale to assess activity ranging from 1 to 10. The patient indicates her or his most appropriate activity level, with 1 defined as ''wholly inactive and dependent on others'' and 10 defined as ''regular participation in impact sports.''
knee injury and osteoarthritis outcome score (KOOS) | 1 month preoperative
  Questionnaire to assess knee outcomes: Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL).
  A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
knee injury and osteoarthritis outcome score (KOOS) | 1 year post-operative
  Questionnaire to assess knee outcomes: Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL).
  A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
knee injury and osteoarthritis outcome score (KOOS) | 2 years post-operative
  Questionnaire to assess knee outcomes: Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL).
  A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Forgotten Joint Score | 1 month preoperative
  Scale that shows how aware patients are of their artificial hip/knee joint in everyday life. Total score range: 0 to 100. Finally, the score is subtracted from 100, to change the direction of the final score in a way that high scores indicate a high degree of "forgetting" the artificial joint, that is, a low degree of awareness.
Forgotten Joint Score | 1 year post-operative
  Scale that shows how aware patients are of their artificial hip/knee joint in everyday life. Total score range: 0 to 100. Finally, the score is subtracted from 100, to change the direction of the final score in a way that high scores indicate a high degree of "forgetting" the artificial joint, that is, a low degree of awareness.
Forgotten Joint Score | 2 years post-operative
  Scale that shows how aware patients are of their artificial hip/knee joint in everyday life. Total score range: 0 to 100. Finally, the score is subtracted from 100, to change the direction of the final score in a way that high scores indicate a high degree of "forgetting" the artificial joint, that is, a low degree of awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Edmonton Bone and Joint Centre, Edmonton, Alberta, Canada